CLINICAL TRIAL: NCT02520401
Title: The Use of a Probiotic Lozenge in the Treatment of Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: s57668
Record Dates: First submitted 2015-05-06; First posted 2015-08-11 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2018-01

CONDITIONS: Peri-implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Test (Experimental): Probiotic tablet
  Interventions: Other: Probiotic - BioGaia
- Control (Placebo Comparator): Control tablet
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Probiotic - BioGaia — Use of a probiotic tablet
  Arms: Test
Other: Placebo — Use of a placebo tablet
  Arms: Control

SUMMARY:
This studies aims to investigate the effect of a probiotics in peri-implantitis patients as an adjunct to non-surgical therapy.

DETAILED DESCRIPTION:
This studies aims to investigate the effect of a probiotics in peri-implantitis patients as an adjunct to non-surgical therapy.

Study design: This study will be a single centre (Department of Oral Health Sciences, University Hospitals Leuven), double blind randomized, placebo controlled clinical trial. The randomization (by means of a computer program) and double blind design are thought to minimize the bias of the investigator and patients.

Selection of the study population: Adults, who consult at the departement of Periodontology at the University Hospital Leuven, with peri-implantitis and who fit the inclusion criteria will be asked to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Patients with at least one implant* diagnosed with initial peri-implantitis.
* Willing and able to give written informed consent
* No signs of acute periodontitis
* presence of keratinized tissue around treated implant(s)

Exclusion Criteria:

* patients who smoke
* patients with periodontitis
* pregnant or lactating woman
* patients with poorly controlled diabetes
* patients taking bisphosphonate mediation
* patient who had taken systemic antibiotics 3 months prior to treatment
* peri-implantitis treatment 12 months prior intake

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth (PPD) at peri-implantitis sites | Baseline - 6 months
  Pocket probing depth measured with Merrit-B probe

SECONDARY OUTCOMES:
Bleeding on Probing (BoP) at peri-implantitis sites | Baseline - 6 months
  Binairy outcome: 0: no bleeding, 1: bleeding
Plaque at peri-implantitis sites | Baseline - 6 months
  Binairy outcome: 0: no plaque, 1: plaque
Microbial samples | Baseline - 6 months
  Of tongue coating, saliva and peri-implantitis site
Full mouth plaque score (FMPS) | Baseline - 6 months
  Binairy outcome: 0: no plaque, 1: plaque

CONTACTS AND LOCATIONS:
Locations (1):
- UZLeuven, Leuven, Belgium